CLINICAL TRIAL: NCT04387643
Title: Protecting Health Care Workers During the COVID-19 Outbreak:Qualitative Study of AYUSH Initiative
Brief Title: Protecting Health Care Workers During the COVID-19 Outbreak
Status: Completed | Type: Observational
Sponsor: Aarogyam UK (Other)
Collaborators: Samta Ayurveda Prakoshtha, India (Unknown)
Responsible Party: Sponsor
Other Study IDs: AU/SA/01
Record Dates: First submitted 2020-05-13; First posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Ayurvedic Kadha — Kadha (also called Kwath and Kashaya) is a type of ayurvedic formulation prepared by boiling herbs in water. Water and herbs are main ingredients of these preparations. The preparation of Kadha uses dry herbs, which are dried under the sun or in the shade, as directed for the individual herb. Then, the herbs are pounded to form a coarse powder

SUMMARY:
Preparing to deal with Covid-19 outbreak in Rajasthan, India, health care workers were given Ayurvedic Kadha (combination of ayurvedic herbal extracts) starting from the end of February 2020. Then, majority of these health care workers were put on front line managing screening, monitoring, quarantine and treating Covid 19 patients. This real-life study aimed to determine the experience of health care workers who had Ayurveda kadha before starting as front-line workers.

ELIGIBILITY:
Inclusion Criteria:

* Health care workers posted in Covid-19 duties at front line
* Health workers who had Ayurveda herbs combination over for at least 10-days

Exclusion Criteria:

* No willing to consent
* inability to participate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Health care workers at front line of Covid-19 screening, treatment and management
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-02 (Actual)

PRIMARY OUTCOMES:
Physical Health | From baseline to 30-days
  Self-reported health issues
Psychological Health | From baseline to 30-days
  Self-reported psychological issues

SECONDARY OUTCOMES:
Coping with distress | From baseline to 30-days
  Self-reported coping with high demanding work in Covid-19 duties
Self-Help | From baseline to 30-days
  Self reported self-help measures used

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, Study Chair — British Ayurvedic Medical Council (UK); Jaydeep Joshi, Study Director — Aarogyam UK; Parashar Sharma, Study Director — Samta Ayurveda Prakoshtha, India; Sahil Singhal, Principal Investigator — Samta Ayurveda Prakoshtha, India
Locations (1):
- Samta Ayurveda Prakoshtha, Jaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: Undecided